CLINICAL TRIAL: NCT01285687
Title: Acupuncture for Post-tonsillectomy Pain Control in Children: a Single-blinded, Randomized, Controlled Study
Brief Title: Acupuncture for Post-tonsillectomy Pain Control in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0076-09-ZIV
Record Dates: First submitted 2011-01-23; First posted 2011-01-28 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Tonsillectomy; Post-Operative Pain; Acupuncture
Keywords: Tonsillectomy; Post-Operative Pain; Acupuncture
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Analgesic Treatment (No Intervention)
- Standard Analgesic Treatment with Acupuncture (Experimental): Patients will receive standard analgesic treatment and in addition acupuncture.
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — Sterile, disposable, FDA-approved acupuncture needles will be used. Acupuncture will be performed bilaterally. The needles will penetrate the skin to a depth of 5-10mm and will be kept in place for no more than 5 minutes. The acupuncture points will be: Li 4, Li 11, St 44, according to Chinese acupuncture mapping. Treatment will be repeated at least 3 times during the hospital stay. Treatment will start in the pediatrics department approximately two hours after discharge from the postoperative unit. The 2nd treatment will be given on the same evening, approximately 4-8 hours after the 1st treatment and the 3rd treatment will be given the following morning, approximately 12-18 hours after the 2nd treatment. Exact treatment times will be recorded in the patient's file.
  Arms: Standard Analgesic Treatment with Acupuncture

SUMMARY:
A randomized, controlled, single-blinded study comparing conventional postoperative analgesia with paracetamol-on-demand with the same regime plus acupuncture.

The hypothesis is that postoperative treatment of children undergoing tonsillectomy with acupuncture will reduce pain with minimal unwanted effects.

DETAILED DESCRIPTION:
A randomized, controlled, single-blinded study comparing conventional postoperative analgesia with paracetamol-on-demand with the same regime plus acupuncture.

The study will be conducted in accordance with the ethical standards of the Helsinki Declaration and has been approved by the Human Experimentation Ethics Committee of the Ziv Medical Center and the Ministry of Health.

Patients will be recruited through the preoperative clinic conducted on the day before surgery. All parents and children will be given a full explanation of the study by an experienced member of the research team before randomization. The explanation will include the nature of acupuncture and the proposed treatment. Parents will sign an informed consent. Patients randomized to the acupuncture group will have a "trial run" at the time of consenting with a member of the research team experienced with performing acupuncture in children , in order to familiarize the child and family with the procedure.

ELIGIBILITY:
Inclusion Criteria:

• children aged 3-12 years undergoing tonsillectomy with or without adenoidectomy for tonsillar hypertrophy with suspected sleep disordered breathing and for recurrent tonsillar infections.

Exclusion Criteria:

* lack of parental consent
* skin lesions near acupuncture sites
* relevant psychiatric disorder
* coagulopathy
* drug allergies to regular analgesic treatment
* intake of medications possibly affecting postoperative pain
* any child who has received acupuncture treatment in the past or the parents or siblings have received such treatment.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Post-Operative Pain | 48 hours post-surgery

SECONDARY OUTCOMES:
Analgesic Drug Consumption | 48 hours post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel